CLINICAL TRIAL: NCT00006213
Title: Phase I Study of Farnesyl Transferase Inhibitor BMS-214662 (NSC 710086) in Acute Leukemias, Myelodysplastic Syndromes (RAEB and RAEB-T) and Chronic Myeloid Leukemia in Blast Phase
Brief Title: BMS-214662 in Treating Patients With Acute Leukemia, Myelodysplastic Syndrome, or Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02338; DM99-290; U01CA062461 (NIH); CDR0000067887 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-09-11; First posted 2003-12-24 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Promyelocytic Leukemia (M3); Blastic Phase Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — 7-cyano-2,3,4,5-tetrahydro-1-(1H-imidazol-4-ylmethyl)-3-(phenylmethyl)-4-(2-thienylsulfonyl)-1H-1,4-benzodiazepine

ARMS (1):
- Treatment (BMS-214662) (Experimental): Patients receive BMS-214662 IV over 1 hour weekly for 4 weeks. Treatment continues every 4 weeks for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: BMS-214662; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: BMS-214662 — Given IV
  Other Names: farnesyltransferase inhibitor BMS-214662; FTI BMS 214662
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Phase I trial to study the effectiveness of BMS-214662 in treating patients who have acute leukemia, myelodysplastic syndrome, or chronic myeloid leukemia in blast phase

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and dose limiting toxicity of BMS-214662 in patients with acute leukemia, myelodysplastic syndrome, or chronic myeloid leukemia in blast phase.

II. Determine any preliminary evidence of antileukemia activity of this drug in these patients.

OUTLINE: This is a dose escalation study.

Patients receive BMS-214662 IV over 1 hour weekly for 4 weeks. Treatment continues every 4 weeks for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of BMS-214662 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have:

  * AML, ALL, or high-risk MDS (RAEB or RAEB-t) that has:

    * Not responded (no CR) to initial induction chemotherapy, or
    * Recurred after an initial CR of < 1 year, or
    * Recurred after an initial CR of > 1 year and failed to respond to an initial reinduction attempt, or
    * Recurred more than once, or
  * Chronic myeloid leukemia in myeloid blast phase

    * Patients with CML blast phase may receive BMS-214662 as their first therapy for blast phase or after failing other treatments for blast phase
  * Patients with refractory or relapsed acute promyelocytic leukemia are eligible provided they have failed an ATRA-containing regimen
* Performance status of =< 0-2
* Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of the hospital
* Patients must have been off chemotherapy for the 4 weeks prior to entering this study and recovered from the toxic effects of that therapy; patients with evidence of rapidly progressive disease (i.e., absolute peripheral blood blast count >= 5 x 10^9/L and increasing by >= 1 x 10^9/L/24 hours) may receive treatment before 4 weeks from the previous treatment providing they have recovered from all toxic effects of that therapy; use of hydroxyurea on patients with rapidly proliferative disease is allowed up to 24 hours prior to the start of therapy
* Bilirubin =< 1.5 mg/dL
* Creatinine =< 1.5 mg/dL or creatinine clearance >= 60 mL/hr
* Patients who are likely to benefit from allogeneic bone marrow transplantation (i.e., age < 60 years of physiological age with histocompatible donor) should be excluded from this study unless such therapy is not feasible

Exclusion Criteria:

* Pregnant and nursing females will be excluded; patients of childbearing potential should practice effective methods of contraception
* Patients with prolonged QTc interval on EKG are excluded

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-04; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which 2 of 6 patients experience DLT assessed using NCI CTC version 2.0 | 4 weeks
  Non-parametric tests will be used to study the relationship between baseline and post-therapy values at different dose levels and times.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States